CLINICAL TRIAL: NCT05764005
Title: Optimizing Active Surveillance in Low-Risk Prostate Cancer: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2022.059; HUM00209599 (Other: University of Michigan); 5K08CA245237 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: low-risk; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention website (Experimental)
  Interventions: Behavioral: web-based tool (MAP- Management of Active surveillance in Prostate Cancer)
- Control MUSIC website (Active Comparator): This is usual care and all urologists are encouraged to refer their patients to the patient educational materials on the MUSIC website (http://www.musicurology.com/patientmaterials/).
  Interventions: Behavioral: MUSIC website

INTERVENTIONS:
Behavioral: web-based tool (MAP- Management of Active surveillance in Prostate Cancer) — A web-based tool with modules on active surveillance education, team based active surveillance care delivery and the role of the PCP, and self-management for cancer anxiety and worry. {may need more detail}
  Arms: Intervention website
Behavioral: MUSIC website — Standard of care educational materials {add more detail}
  Arms: Control MUSIC website

SUMMARY:
This is a pilot evaluation of a patient-centered intervention that enables providers to support men on active surveillance to maximize adherence. Conducted in urology practices, this pilot will measure key patient-reported, provider-reported, and implementation outcomes. Successful completion of this work will inform a subsequent multi-center effectiveness-implementation hybrid design trial and ultimately will improve low-risk cancer management by effectively engaging Primary Care Physicians (PCPs) in care delivery.

ELIGIBILITY:
Patient Inclusion Criteria:

* 55 years old or older
* Men diagnosed with low-risk prostate cancer currently on active surveillance
* Men who identify having a primary care provider
* Access and ability to use the Internet

Patient Exclusion Criteria:

* Men who are unable to read and/or speak English
* Men with impaired decision-making capacity (such as with a diagnosis of dementia or memory loss)

PCP Inclusion Criteria:

* Identified by patient on baseline survey as their PCP

Urologist and Clinic Staff Inclusion Criteria:

* Clinicians or staff at a participating urology clinic, including but not limited to MDs, APPs, and nurses

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Feasibility - recruitment | up to 9 months post last patient recruitment
  Defined as the successful recruitment of 40 patients.
Feasibility - Uptake | up to 6 months post last patient recruitment
  Defined as the proportion of men who complete the baseline and follow-up surveys out of the total number of patients recruited.
Acceptability - Mean Satisfaction Scores | up to 4 months post last patient completing intervention
  Acceptability asks the extent to which participants consider the intervention is agreeable. Patients in the intervention arm will answer questions (on a 5-point Likert scale) regarding the use of the tool including: a) the tool provided me the necessary information about being on active surveillance; b) the tool helped me know what tests I needed and when; c) the tool helped me understand what my PCP can do for my active surveillance; d) the tool was easy to use; e) the amount of time it took to go through the website; and f) I would recommend the tool to other patients. We will ask an open-ended question on if the tool should have any other features in future versions. We will additionally collect paradata such as user actions (clicks) and time spent on each webpage.

CONTACTS AND LOCATIONS:
Overall Officials: Archana Radhakrishnan, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided